CLINICAL TRIAL: NCT03942991
Title: Anesthetic Efficacy Of 4% ArtpharmaDent Versus 2% Mepecaine-L for Infilteration Anesthesia in Extraction of Badly Decayed Lower First Primary Molars: Pilot Study
Brief Title: Anesthetic Efficacy Of 4% ArtpharmaDent Versus 2% Mepecaine-L in Extraction of Lower First Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadeen Hossam Eldin Hosny Ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14422017496941
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Badly Decayed Lower First Primary Molars in Children
MeSH Terms: interventions — Carticaine; Mepivacaine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% Mepecaine-L (Active Comparator): infiltration injection of 2% Mepivacaine
  Interventions: Drug: Mepivacaine 2% Injection
- 4% Artpharmadent (Experimental): infiltration injection of 4% Articaine
  Interventions: Drug: articaine

INTERVENTIONS:
Drug: articaine — infiltration injection of 4%artpharmadent
  Other Names: Artpharmadent
  Arms: 4% Artpharmadent
Drug: Mepivacaine 2% Injection — infiltration injection of 2% Mepecaine-L
  Other Names: 2% Mepecaine-L
  Arms: 2% Mepecaine-L

SUMMARY:
parallel technique will be done where the investigator (will be blinded) will give one type on anesthesia then performing the extraction and evaluating the intraoperative pain ,the same procedure will be done for the other type of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-8 years.
* Medically fit (ASA I, II).
* Mentally capable of communication.
* Having a mandibular first primary molar tooth that require Extraction.
* Child must give assent prior to participation, as well as parental informed written consent.
* Body weight >20 kg.
* it should be the first dental treatment to the child

Exclusion Criteria:

* Medically and mentally compromised children.
* Children without a history of prolonged bleeding, platelet disorders, hypersensitivity,
* History of significant behavior management problems.
* Patients having active sites of pathosis in the area of injection.
* Patients who had taken analgesics or antibiotics in the 12-hrs preceding the injection.
* Patients allergic to Articaine and/or Mepivacaine and/or sulfur

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Intra-Operative Pain during Extraction | Immediatly after etxraction
  intraoperative pain will be measured using wong baker pain scale,The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain Face